CLINICAL TRIAL: NCT02989038
Title: Reactions to Reduced Nicotine Cigarettes in Young Adult Low-Frequency Smokers
Acronym: NicRed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00075882; R01DA042532 (NIH)
Record Dates: First submitted 2016-09-23; First posted 2016-12-12 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Nicotine Dependence
Keywords: smoker; young adult; adolescent
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Products

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- NNC, INC, VLNC (Experimental): Normal Nicotine Content (NNC), Intermediate Nicotine Content (INC), Very Low Nicotine Content (VLNC)
  Interventions: Other: Very Low Nicotine Content Cigarettes; Other: Intermediate Nicotine Content Cigarettes; Other: Normal Nicotine Content Cigarettes
- NNC, VLNC, INC (Experimental): Normal Nicotine Content, Very Low Nicotine Content, Intermediate Nicotine Content
  Interventions: Other: Very Low Nicotine Content Cigarettes; Other: Intermediate Nicotine Content Cigarettes; Other: Normal Nicotine Content Cigarettes
- INC, VLNC, NNC (Experimental): Intermediate Nicotine Content, Very Low Nicotine Content, Normal Nicotine Content
  Interventions: Other: Very Low Nicotine Content Cigarettes; Other: Intermediate Nicotine Content Cigarettes; Other: Normal Nicotine Content Cigarettes
- INC, NNC, VLNC (Experimental): Intermediate Nicotine Content, Normal Nicotine Content, Very Low Nicotine Content
  Interventions: Other: Very Low Nicotine Content Cigarettes; Other: Intermediate Nicotine Content Cigarettes; Other: Normal Nicotine Content Cigarettes
- VLNC, NNC, INC (Experimental): Very Low Nicotine Content, Normal Nicotine Content, Intermediate Nicotine Content
  Interventions: Other: Very Low Nicotine Content Cigarettes; Other: Intermediate Nicotine Content Cigarettes; Other: Normal Nicotine Content Cigarettes
- VLNC, INC, NNC (Experimental): Very Low Nicotine Content, Intermediate Nicotine Content, Normal Nicotine Content
  Interventions: Other: Very Low Nicotine Content Cigarettes; Other: Intermediate Nicotine Content Cigarettes; Other: Normal Nicotine Content Cigarettes

INTERVENTIONS:
Other: Very Low Nicotine Content Cigarettes — cigarettes with 0.03 nicotine yield with 0.4 mg/g nicotine content and 9.0 mg tar yield
  Other Names: Tobacco; Cigarettes
Other: Intermediate Nicotine Content Cigarettes — cigarettes with 0.12 nicotine yield with 2.4 mg/g nicotine content and 9.0 mg tar yield
  Other Names: Tobacco; Cigarettes
Other: Normal Nicotine Content Cigarettes — cigarettes with 0.8 nicotine yield with 15.8 mg/g nicotine content and 10.5 mg tar yield
  Other Names: Tobacco; Cigarettes

SUMMARY:
The purpose of this study is to evaluate reactions to, and choices to self-administer, cigarette smoke with varying nicotine content among low-frequency, non-dependent adolescent/young adult smokers between the ages of 15-25 years.

DETAILED DESCRIPTION:
Participants will undergo three sessions in which their reactions to fixed doses of smoke from investigational cigarettes with three different nicotine contents (15.8 mg/gram of tobacco, 2.5 mg/g, and .4 mg/g) will be assessed. Following the third fixed-dose session, participants will return to the lab to choose one of the cigarettes to self-administer.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* between the ages of 15-25
* use nicotine or tobacco products between 1-15 days/month for at least 6 months
* smokes at least 5 cigarettes/month
* no unstable or significant medical or psychiatric conditions
* breath alcohol value=0.000
* able to provide contact information for two individuals who can corroborate smoking status

Exclusion Criteria:

* use of illegal drugs as measured by urine drug screen (excluding THC)
* serious quit attempt in the past 3 months
* plans to quit smoking in the next 2 months
* current use of nicotine replacement therapy or other tobacco cessation products
* inability to attend all required experimental sessions
* blood pressure >160/100 mmHg
* pregnant, trying to become pregnant, or breastfeeding

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Subjective reactions to fixed doses of tobacco smoke | Immediately after puff administration of each study cigarette
  Smoking Effects Questionnaire ratings following administration of puffs for NNC, INC, and VLNC cigarettes
Cigarette choice | 30 minutes after sampling all 3 study cigarettes
  Participants will choose which of the three cigarettes they prefer to smoke by ranking each of the three cigarette conditions using a 1-3 scale where 1 is the cigarette that they most desire to smoke and 3 is the cigarette that they least desire to smoke.

SECONDARY OUTCOMES:
Mood and Affect | Immediately after puff administration of each study cigarette
  The Positive and Negative Affect Schedule (PANAS)
Mood and Affect | Immediately after puff administration of each study cigarette
  Minnesota Nicotine Withdrawal Scale (MNWS)
Smoking topography - Change in Carbon Monoxide (CO) values (in parts per million, ppm) following puff administration | Immediately after puff administration of each study cigarette
  CO values (in ppm) will be obtained using a handheld CO monitor prior to puff administration and 5 minutes after completion of cigarette puff administration. The difference in values will provide a CO boost value
Smoking topography - number of puffs | During self-administration of chosen cigarette at the last experimental session (approximately over 10 minutes)
  number of puffs
Smoking topography - interpuff interval | During self-administration of chosen cigarette at the last experimental session (approximately over 10 minutes)
  Interpuff interval (in seconds) will be calculated using video recordings of self-administration of chosen cigarette

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No